CLINICAL TRIAL: NCT05095142
Title: Preventive and Personalized Medicine (2021-2023)
Brief Title: The Role of Genetic Factors in the Development of Idiopathic Osteoarthritis of the Knee in the Kazakh Population
Status: Completed | Type: Observational
Sponsor: Asfendiyarov Kazakh National Medical University (Other)
Responsible Party: Principal Investigator, Ildar Fakhradiyev, Head of the Laboratory of Experimental Medicine, Asfendiyarov Kazakh National Medical University
Other Study IDs: 1191
Record Dates: First submitted 2021-10-21; First posted 2021-10-27 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Idiopathic Osteoarthritis
Keywords: SNP

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group:: patients with idiopathic osteoarthritis of the knee
  Interventions: Genetic: SNP analysis of the DNA
- Control group: patients without idiopathic osteoarthritis of the knee
  Interventions: Genetic: SNP analysis of the DNA

INTERVENTIONS:
Genetic: SNP analysis of the DNA — SNP analysis of the DNA obtained from peripheral blood sample

SUMMARY:
The purpose of this study is to identify genetic determinants of susceptibility to idiopathic osteoarthritis of the knee . It will assist in predicting individual risks of disease progression and would help to clarify pathophysiologic mechanisms of idiopathic osteoarthritis of the knee

ELIGIBILITY:
Inclusion Criteria:

1. Patients with bilateral idiopathic gonarthrosis aged 18 to 65 years;
2. Representatives of the Kazakh ethnic group up to the 3rd generation;
3. Hereditary history of arthrosis;
4. Persons who are able and willing to provide written informed consent;

Exclusion Criteria:

1. Patients with bilateral idiopathic gonarthrosis under 18 years of age and over 65 years of age;
2. Representatives of other ethnic groups;
3. Representatives of the Kazakh ethnic group less than 3 generations;
4. No family history of bilateral idiopathic gonarthrosis;
5. Patients with an acute period of the inflammatory process (laboratory and clinical signs);
6. Persons who, in the opinion of the researcher, are mentally or legally incapacitated, which prevents obtaining informed consent;
7. Pregnant or lactating women;
8. Tuberculosis of any localization in the active phase and in history;
9. Severe and decompensated diseases of the liver and kidneys, cardiovascular system;
10. Severe and decompensated course of endocrine diseases;
11. Autoimmune diseases;
12. Systemic diseases;
13. Oncological diseases;

Ages: 18 Years to 68 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Persons of Kazakh nationality
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
enotyping for the SNP associated with liver cirrhosis | 1 year
  Genotype frequency of SNP in the study genes of participants and control participants.

CONTACTS AND LOCATIONS:
Overall Officials: Olzhas Bekarisov, PhD, Principal Investigator — Scientific center of traumatology and orthopedics named after academician Batpenova ND
Locations (1):
- Scientific center of traumatology and orthopedics named after academician Batpenova ND, Almaty, Kazakhstan